CLINICAL TRIAL: NCT02176213
Title: A Phase II Study of Pomalidomide, Daily Low Dose Oral Cyclophosphamide, and Dexamethasone in Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Pomalidomide, Cyclophosphamide, Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajai Chari (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Ajai Chari, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-0825; PO-CL-MM-PI-002404
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Relapsed; Refractory; Multiple Myeloma; Pomalidomide; Cyclophosphamide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomalidomide, Cyclophosphamide, Dexamethasone (Experimental): Three oral drugs will be given in 28-day cycles: Pomalidomide 4 mg daily x 21 days; cyclophosphamide 50 mg BID x 21 days; and dexamethasone 40 mg weekly x 3 (20 mg weekly if the patient aged ≥ 75 years old)
  Interventions: Drug: Pomalidomide; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — 4 mg PO x 21 days
  Other Names: pomalyst
Drug: Cyclophosphamide — low dose cyclophosphamide 50 mg PO BID x 21 days
  Other Names: cytoxan
Drug: Dexamethasone — dexamethasone 40 mg PO weekly (or 20 mg if ≥ 75 years old).

SUMMARY:
This study is being done to learn more about the drug, pomalidomide and to gather data on its safety and side effects when used in combination with commercially available cyclophosphamide and dexamethasone. This combination is considered experimental and has not been approved by the FDA.

Pomalidomide is a third generation immunomodulatory (IMiDs) agent, which is a more potent version of thalidomide and lenalidomide drugs that have been approved by the United States Food and Drug Administration [FDA] for the treatment of MM. In February 2013, pomalidomide was also approved by the FDA for patients with MM who have had more than 2 types of therapy.

Pomalidomide is taken orally as capsules, and cyclophosphamide and dexamethasone are also taken orally as tablets in this study. Cyclophosphamide and dexamethasone are commercially available and are often used in combination with other drugs to treat Multiple Myeloma. Preliminary data from both the laboratory and patient studies suggest that this combination of drugs is more effective than pomalidomide and dexamethasone alone. However, the regimen being used in this study, which consists of daily cyclophosphamide, also permits support of low blood counts with either injections or transfusions as needed.

DETAILED DESCRIPTION:
This is an open label, single center, phase II study of a combination of pomalidomide, daily low dose oral cyclophosphamide, and dexamethasone in patients with relapsed/refractory multiple myeloma. The three oral drugs will be given in 28-day cycles: Pomalidomide 4 mg daily x 21 days; cyclophosphamide 50 mg BID x 21 days; and dexamethasone 40 mg weekly x 3 (20 mg weekly if the patient aged ≥ 75 years old). Subjects meeting eligibility criteria with ANC < 1000/µL and platelet count < 50,000/µL will start at dose level -1 of both pomalidomide (3 mg daily) and cyclophosphamide (50 mg daily). G-CSF and platelet transfusion support is permitted if needed.

Dose reduction for hematologic toxicity will begin with cyclophosphamide and then subsequently alternate with pomalidomide until a subject cannot tolerate dose level -2 of both agents - in which case subject would come off study. If subject has 2 or more concurrent toxicities that are potentially attributable to both agents (e.g. hematologic toxicity) then dose modification guidelines will be followed with dose reduction being done sequentially with one agent at a time, unless in the opinion of the investigator, both agents required concurrent dose reduction.

ELIGIBILITY:
Inclusion Criteria:

Disease related:

* Patients must have a history of symptomatic multiple myeloma according to the IMWG criteria
* Patients must have received at least two prior lines of therapy and also must be refractory to lenalidomide.
* Patient has relapsed or relapsed/refractory MM.
* Patients must currently have measurable disease, as defined as:

  1. Serum M-protein ≥ 0.5 g/dL
  2. Urine M-protein ≥ 200 mg/24 hours
  3. Serum free light chain assay: involved FLC level ≥ 10 mg/dl provided serum FLC ratio is abnormal
  4. If no monoclonal protein is detected, then > 30% monoclonal bone marrow plasma cells

Demographic:

* Male or female adults ≥ 18 years old
* Able to sign informed consent and to comply with the protocol
* Life expectancy > 12 weeks
* ECOG performance status ≤ 2
* All study participants must be registered into the mandatory POMALYST REMS program, and be willing and able to comply with the requirements of the POMALYST REMS program.

Laboratory

* ANC ≥ 1000/µL
* Platelets ≥ 50,000/µL (Patients with plasma cells 50% of bone marrow nucleated cells, and platelets ≥ 30,000/µL will be permitted regardless of the baseline ANC)
* Cr < 3
* AST ≤ 2.5 x ULN
* ALT ≤ 2.5 x ULN
* Serum Bilirubin ≤ 1.5 x ULN (except patients with Gilbert's syndrome who must have a total bilirubin of <3 time ULN)

Other

* Females of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control at least 28 days before taking pomalidomide.

Exclusion Criteria:

* Previous treatment with pomalidomide
* Patients who received chemotherapy or radiation therapy to 30% of marrow-bearing bone within ≤ 2 weeks or experimental agent/therapy within 4 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide or similar drugs
* Other concurrent severe and/or uncontrolled medical conditions including abnormal laboratory values that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients for whom prophylactic anticoagulation therapy is not an option unless due to thrombocytopenia
* Patients who received allogenic stem cell transplantation < 12 months prior to entering the study or show evidence of active graft-versus-host disease that requires immunosuppressive therapy
* Patients with existing peripheral neuropathy grade > 2
* Patients with an active malignancy requiring treatment in the next 12 months (except for basal or squamous cell carcinoma, or in situ cancer of the cervix or breast, and asymptomatic prostate cancer)
* Patients with known positivity for HIV or active hepatitis B or C
* Corticosteroid therapies of > 20 mg/day prednisone, > 4 mg/day dexamethasone, > 80 mg/day hydrocortisone, or equivalent. Oral, inhaled, or topical steroids are allowed during study as long as it does not exceed 80 mg/day hydrocortisone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Best overall response rate (ORR) | up to 24 months
  disease response

SECONDARY OUTCOMES:
Stringent complete response (sCR) | up to 24 months
Complete response (CR) | up to 24 months
Very good partial response (VGPR) | up to 24 months
Partial response (PR) | up to 24 months
Time to progression (TTP) | up to 24 months
  TTP is defined as beginning with the time the first dose of PCD regimen is administered until disease progression on PCD regimen.
Duration of response (DOR) | up to 24 months
  DOR is defined as the time from first evidence of PR or better to confirmation of disease progression.
Clinical benefit response (CBR) | up to 24 months
  CBR is the combination of the ORR and minimal response (MR) i.e. this includes sCR, CR, VGPR, PR, and MR.
Progression free survival (PFS) | up to 24 months
  PFS is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier.
Overall survival (OS) | up to 24 months
  OS is defined as the time from the first dose of study treatment to the date of death (whatever the cause).

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Chari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States